CLINICAL TRIAL: NCT05427422
Title: Motor Recovery of Stroke Patients Based on Electroencephalogram-functional Magnetic Resonance Imaging
Brief Title: Stroke Recovery Research Based on EEG-fMRI
Acronym: EEG-fMRI
Status: Completed | Type: Observational
Sponsor: Xi'an Jiaotong University (Other)
Collaborators: Xian Daxing Hospital (Unknown)
Responsible Party: Principal Investigator, Wentao Zeng, PhD candidate, Xi'an Jiaotong University
Other Study IDs: Stroke01
Record Dates: First submitted 2022-06-14; First posted 2022-06-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Motor Neuropathy
Keywords: motor function recovery; ischemic stroke; EEG-fMRI; neural plasticity
MeSH Terms: conditions — Neuritis; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- High Recovery: Effective recovery rate defined as difference between Fugl-meyer scores in the 6 weeks after stroke onset (eF) and in the enrollment (sF) normalized by (total score-sf) would be used to indicate the recovery Level of a patients, i.e., (eF-sF)/ (total score-sf). A previously reported recovery rate, i.e., proportional recovery((eF-sF)/(total score-sf)=0.7) was chosen as a standard of a high recovery. Patients with effective recovery rate higher than 0.7 at the T1 time point (6 weeks after stroke onset) would be assigned to group with high recovery rate
  Interventions: Diagnostic Test: MRI recording; Diagnostic Test: EEG recording
- Low Recovery: The Low Recovery group indicates that patients with effective recovery rate lower than 0.7
  Interventions: Diagnostic Test: MRI recording; Diagnostic Test: EEG recording
- Healthy Control: Age/sex matched healthy subjects enrolled to compare with group of patients.
  Interventions: Diagnostic Test: MRI recording; Diagnostic Test: EEG recording

INTERVENTIONS:
Diagnostic Test: MRI recording — MRI imaging was performed using a 3 Tesla Siemens Prisma system with a 64-channel head/neck coil (Siemens Medical Systems, Erlangen, Germany). The MRI protocols included as follows: (i) Magnetization-Prepared 2 Rapid Acquisition Gradient Echoes: TR/TE/ TI1/TI2 = 5000/2.98/700/2500 ms, voxel size = 1.0 × 1.0 × 1.0 mm3, FOV = 256 × 240 × 176 mm3; (ii)Gradient-echo EPI: TR 720 ms, TE 33.1 ms, flip angle 52 deg, FOV 208x180 mm, Matrix 104x90, Slice thickness 2.0 mm; 72 slices; 2.0 mm isotropic voxels, Multiband factor 8, Echo spacing 0.58 ms, BW 2290 Hz/Px; (iii) DSI : TR/TE = 3300/73 ms, FOV = 220 × 220 × 60 mm3, voxel size = 2 × 2 × 2 mm3, 128 diffusion direction, b-max = 3000 sec/mm2, AT = 7:22 min); (iv) T2-weighted fluid-attenuated inversion recovery: TR/TE = 9000/84 ms, FOV = 270 × 320 × 22 mm2, voxel size = 0.72 × 0.72 × 6.6 mm3.
Diagnostic Test: EEG recording — EEG was performed using a BrainAmp MR 32 amplifier (BrainProducts GmbH, München, Germany). The EEG protocols included as follows: (i) EEG-fMRI fusion: Sampling rate: 5000 Hz, low cut off-high cut off: DC-1000Hz;(2) EEG-fMRI fusion: Sampling rate: 1000 Hz, low cut off-high cut off: DC-1000Hz.
  In (i) an ECG channel would be used to collect artifact of pulse and not used in (ii).

SUMMARY:
This study is aimed to investigate the post-stroke motor recovery of patients with ischemic stroke based on their neural features extracted from EEG-fMRI data.

DETAILED DESCRIPTION:
A group of patients with ischemic stroke and age/gender matched healthy controls would be enrolled in this study. Their features of neural activities based on EEG-fMRI fusion scan would be extracted to investigate the mechanisms of motor recovery after stroke. Particularly, the correlations of their features of neural networks or local activities to their motor function (defined as their Fugl-Meyer scores) at enrollment and their recovery time courses consisted of Fugl-Meyer scores in follow-up time points. Data of T1 structural, DSI fiber image and pure EEG (without MRI) would also be collected along with EEG-fMRI fusion data.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 and below 75 years
* Motor impairment in National Institutes of Health Stroke Scale
* 7-14 days since stroke attack
* First-ever ischemic stroke

Exclusion Criteria:

* Motor impairment induced by non-stroke aetiology
* Claustrophobia; recognition disorder
* History of other severe central nervous system diseases
* Any signs unfit for MRI/EEG scan

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AA population with motor impairment induced by first-ever stroke in a specific duration (7-14 days after stroke attack, i.e., early subacute stage) would be enrolled to investigate the mechanisms of post-stroke recovery of motor function.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer scores (T0) | 7-14 days since stroke
  a scale widely used to evaluate one's motor impairment
Fugl-Meyer scores (T1) | 6 weeks since stroke
  a scale widely used to evaluate one's motor impairment
Fugl-Meyer scores (T2) | 12 weeks since stroke
  a scale widely used to evaluate one's motor impairment
Fugl-Meyer scores (T3) | 72 weeks since stroke
  a scale widely used to evaluate one's motor impairment

SECONDARY OUTCOMES:
Neuroimage features based on EEG-fMRI (T0) | 7-14 days since stroke
  Neuroimage features extracted from EEG-fMRI data
Neuroimage features based on EEG-fMRI (T1) | 6 weeks since stroke
  Neuroimage features extracted from EEG-fMRI data
Neuroimage features based on EEG-fMRI (T2) | 12 weeks since stroke
  Neuroimage features extracted from EEG-fMRI data
Neuroimage features based on EEG-fMRI (T3) | 72 weeks since stroke
  Neuroimage features extracted from EEG-fMRI data

CONTACTS AND LOCATIONS:
Locations (1):
- Xi'an Daxing Hospital, Xi’an, Shanxi, China